CLINICAL TRIAL: NCT04990674
Title: Acute-REMOTION: a Randomized Controlled Pilot Trial to Investigate the Feasibility and Potential Effects of a Transdiagnostic Treatment to Reduce Symptom Severity and Improve Emotion Regulation in Acute Psychiatric Patient Care
Brief Title: Acute-REMOTION: REMOTION in Acute Psychiatric Care
Acronym: Acute-REMOTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01139
Record Dates: First submitted 2021-07-15; First posted 2021-08-04 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REMOTION + TAU (Experimental)
  Interventions: Behavioral: REMOTION; Behavioral: TAU
- TAU (Active Comparator)
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: REMOTION — REMOTION is an internet-based program focusing on emotion regulation and aimed at reducing patient symptom severity and improving emotion regulation. It consists of six modules and the structure is based on the extended process model of emotion regulation by Gross (2015). The intervention is currently being studied in an outpatient psychotherapy setting (Bielinski et al., 2020).
  Arms: REMOTION + TAU
Behavioral: TAU — Treatment as usual (TAU), refers to standard treatment in an acute inpatient care setting at the Universitäre Psychiatrische Dienste Bern. This treatment includes different standard inpatient psychiatric care components (integrative psychiatric care).

SUMMARY:
This study aims to examine REMOTION, an internet-based intervention aimed at reducing symptom severity and improving emotion regulation in an acute psychiatric inpatient care setting. REMOTION is currently being studied in an outpatient psychotherapy setting. This study aims to investigate feasibility and first effects of this intervention in inpatient psychiatric care.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* In acute inpatient care
* With internet access
* Informed consent given

Exclusion Criteria:

* Current participation in another specific emotion regulation intervention group
* Current or history of psychotic disorders, bipolar disorder, mental retardation or organic mental disorders
* Acute suicidality
* Insufficient mastery of German language

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Change in general symptom severity | Assessed at Baseline
  Assessed with the Brief Symptom Inventory 18 (BSI-18)
Change in general symptom severity | Assessed after 4 weeks
  Assessed with the Brief Symptom Inventory 18 (BSI-18)
Change in general symptom severity | Assessed after inpatient discharge (on average 24 days after inpatient intake)
  Assessed with the Brief Symptom Inventory 18 (BSI-18)
Change in general symptom severity | Assessed after 8 weeks
  Assessed with the Brief Symptom Inventory 18 (BSI-18)

SECONDARY OUTCOMES:
Difficulties in emotion regulation | Assessed at Baseline, then after 4 Weeks, after inpatient discharge (on average 24 days after inpatient intake), and after 8 Weeks
  Assessed with the Difficulties in Emotion Regulation Scale (DERS)
Emotion regulation skills | Assessed at Baseline, then after 4 Weeks, after inpatient discharge (on average 24 days after inpatient intake), and after 8 Weeks
  Assessed with the Self-Report Measure for the Assessment of Emotion Regulation Skills (SEK-27)
Usability of REMOTION | Assessed after 4 weeks, after inpatient discharge (on average 24 days after inpatient intake), and after 8 Weeks
  Assessed with the System Usability Scale (SUS)
Satisfaction with REMOTION | Assessed after 4 Weeks, after inpatient discharge (on average 24 days after inpatient intake), and after 8 Weeks
  Assessed with the ZUF-8 (Fragebogen zur Messung der Patientenzufriedenheit) Questionnaire adapted for an internet-based program
REMOTION usage parameters | Assessed after 4 weeks, after inpatient discharge (on average 24 days after inpatient intake) and after 8 weeks
  Amount of modules completed and amount of exercises completed
Qualitative interviews with healthcare workers | 4 months after study start
  Recorded interviews on the topic of attitudes towards / barriers and facilitators / advantages and disadvantages of internet-based interventions in inpatient care
Qualitative interviews with patients lost to follow up | After a patient is lost to follow-up (after the 8 week timepoint when follow-up is assessed, has passed for the individual patient)
  Individuals lost to follow up can take part in a telephone interview on a voluntary basis, this examines reasons for loss to follow up

CONTACTS AND LOCATIONS:
Overall Officials: Franz Moggi, Prof. Dr., Principal Investigator — Universitäre Psychiatrische Dienste Bern, Universität Bern
Locations (1):
- Universitäre Psychiatrische Dienste Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bielinski LL, Walchli G, Lange A, von Kanel E, Demel LK, Nissen C, Moggi F, Berger T. A qualitative analysis of healthcare professionals' experiences with an internet-based emotion regulation intervention added to acute psychiatric inpatient care. BMC Psychiatry. 2024 Dec 27;24(1):955. doi: 10.1186/s12888-024-06365-z. PMID 39731056
- [Derived] Bielinski LL, Walchli G, Nissen C, Berger T, Moggi F. Does an Internet-Based Emotion Regulation Intervention Provide Added Value for Acute Psychiatric Inpatient Care? Protocol for a Randomized Controlled Pilot Trial. JMIR Res Protoc. 2023 Jul 11;12:e47656. doi: 10.2196/47656. PMID 37432724